CLINICAL TRIAL: NCT00402051
Title: A Randomized Phase 2 Study of Pemetrexed in Combination With Cisplatin or Carboplatin in the First Line Therapy of Advanced NSCLC
Brief Title: Chemotherapy With Pemetrexed in Combination With Platinum for Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11077; H3E-SB-S109 (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-11-17; First posted 2006-11-22 (Estimated); Results first posted 2010-01-07 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pemetrexed + Cisplatin (Experimental)
  Interventions: Drug: Pemetrexed; Drug: Cisplatin
- Pemetrexed + Carboplatin (Experimental)
  Interventions: Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Drug: Pemetrexed — 500 mg/m2, intravenous (IV), every 21 days x 6 cycles
  Other Names: LY231514; Alimta
Drug: Cisplatin — 75 mg/m2, intravenous (IV), every 21 days x 6 cycles
  Arms: Pemetrexed + Cisplatin
Drug: Carboplatin — Area under the concentration curve (AUC) 5, intravenous (IV), every 21 days x 6 cycles
  Arms: Pemetrexed + Carboplatin

SUMMARY:
This is a two-arm, parallel, open-label, Phase 2 multicenter study of pemetrexed as first line combination therapy with either cisplatin or carboplatin in the palliative setting of stage IIIb and IV non-small cell lung cancer patients. Approximately 130 patients will be included in about 15 centers in Germany and randomized to one of the above treatment regimens in a 1:1 ratio. Chemotherapy will be administered over a maximum of six cycles with a standard length of 21 days. Primary objective will be the Progression Free Survival Time of patients as assessed in both treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically and/or histologically confirmed NSCLC Stage IIIb or IV
* No previous systemic chemotherapy for this cancer
* At least one uni-dimensionally measurable lesion meeting Response Evaluation Criteria In Solid Tumors (RECIST) criteria
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0 or 1 and adequate organ function
* Prior radiation therapy allowed but limited to <25% of the patient's bone marrow

Exclusion Criteria:

* Serious concomitant systemic disorder or active infection
* Mild to moderate renal insufficiency, but unable to interrupt salicylates or other nonsteroidal anti-inflammatory drugs
* Symptomatic central nervous system (CNS) metastases requiring concurrent corticosteroid therapy
* Presence of clinically significant third-space fluid collections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2006-11; Primary Completion 2008-12 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLilly (1-877-285-4559) or 1-317-615-4559 Mon -Fri 9 AM - 5 PM Eastern time (UTC/GMT -5 hours EST), Study Director — Eli Lilly and Company
Locations (12):
- Germany (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coswig
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Großhansdorf
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halle
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hofheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Homburg/Saar
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Immenhausen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lübeck
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., München

REFERENCES:
- [Derived] Schuette WH, Groschel A, Sebastian M, Andreas S, Muller T, Schneller F, Guetz S, Eschbach C, Bohnet S, Leschinger MI, Reck M. A randomized phase II study of pemetrexed in combination with cisplatin or carboplatin as first-line therapy for patients with locally advanced or metastatic non-small-cell lung cancer. Clin Lung Cancer. 2013 May;14(3):215-23. doi: 10.1016/j.cllc.2012.10.001. Epub 2013 Jan 16. PMID 23332288
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 136 patients signed informed consent. Of these, 3 patients were discontinued prior to randomization (1x protocol entry criteria not met, 2x patient decision); 133 patients were randomized, 130 patients started study drug.
Groups:
- Pemetrexed + Cisplatin: Pemetrexed 500 mg/m2 intravenous (IV); Cisplatin 75 mg/m2 IV, every 21 days for 6 cycles
- Pemetrexed + Carboplatin: Pemetrexed 500 mg/m2 intravenous (IV); Carboplatin area under the concentration curve (AUC) 5 IV, every 21 days for 6 cycles
Period: Overall Study
Arm/Group | Pemetrexed + Cisplatin | Pemetrexed + Carboplatin
Started | 66 | 67
Received Treatment | 65 | 65
Completed | 28 (Completed 6 treatment cycles and 30 days of follow-up after last dose of study drug) | 32 (Completed 6 treatment cycles and 30 days of follow-up after last dose of study drug)
Not Completed | 38 | 35
Not completed — Progressive Disease | 13 | 20
Not completed — Adverse Event | 11 | 4
Not completed — Physician Decision | 7 | 3
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Death - Related to Study Drug | 1 | 2
Not completed — Death Due to Study Disease | 2 | 1
Not completed — Death Due to Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pemetrexed + Cisplatin | Pemetrexed + Carboplatin | Total
Number analyzed (Participants) | 65 | 65 | 130
Age Continuous [Mean (Standard Deviation); unit: years] | 62.3 (8.43) | 62.4 (7.51) | 62.4 (7.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 19 | 42
  Male | 42 | 46 | 88
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 65 | 65 | 130
Region of Enrollment [Number; unit: participants]
  Germany | 65 | 65 | 130
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    0 - Fully Active | 40 | 45 | 85
    1 - Ambulatory, Restricted Strenuous Activity | 25 | 20 | 45
Histopathology [Number; unit: participants]
  Squamous Cell Carcinoma | 12 | 13 | 25
  Adenocarcinoma | 38 | 44 | 82
  Large Cell Carcinoma | 6 | 3 | 9
  Mixed Cell Carcinoma | 0 | 1 | 1
  Bronchioalveolar Carcinoma | 0 | 1 | 1
  NSCLC, Not Otherwise Specified | 9 | 3 | 12
Presence of Bone and Brain Metastases [Number; unit: participants] — Presents specifically participants with bone and brain metastases
  participants
    Bone Metastases | 14 | 11 | 25
    Brain Metastases | 2 | 1 | 3
Smoking Status [Number; unit: participants]
  Never Smoked | 9 | 7 | 16
  Past Smoker | 41 | 42 | 83
  Current Smoker | 15 | 16 | 31
Stage of disease [Number; unit: participants] — For all patients randomized, N=66 for Pemetrexed + Cisplatin, N=67 for Pemetrexed + Carboplatin
  participants
    Stage IIIb (locally advanced disease) | 5 | 9 | 14
    Stage IV (metastatic disease) | 61 | 58 | 119
Time Since Patient Stopped Smoking [Mean (Standard Deviation); unit: years] — For past smokers only: N=41 for Pemetrexed + Cisplatin, N=42 for Pemetrexed + Carboplatin
  years | 10.1 (12.31) | 7.4 (10.56) | 8.7 (11.46)
Use of Tobacco Products [Mean (Standard Deviation); unit: years] — For past and current smokers only: N=56 for Pemetrexed +
  Cisplatin, N=58 for Pemetrexed + Carboplatin:
  years | 31.7 (12.74) | 34.6 (11.47) | 33.2 (12.15)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Surviving Progression-Free at 6 Months (Progression Free Survival [PFS] Rate)
Description: For this study, we used the exponential distribution (assumption done for the calculation of the sample size) to estimate the PFS rate. The PFS rate (%) and the 95% confidence intervals were calculated based on the following formula: exp(-6 λ) ± 1.96 * exp(-6 λ) * (-6 λ)/√r. Where λ was calculated based on the Maximum-Likelihood estimator for ln(λ) as given by (Collett 2003): ln(λ) = ln[ r / ∑ti ] with r = number of patients with events up to 6 months, ti = survival time of patient i (i=1,…,n), event or censored up to 6 months, and n= total number of patients per treatment group.
Time Frame: Randomization to Month 6
Population: Full Analysis Set: All patients randomized who received at least one dose of study drug
Measure: Number; unit: percentage
Arm/Group | Pemetrexed + Cisplatin | Pemetrexed + Carboplatin
Number analyzed (Participants) | 65 | 65
percentage | 52.8 [40.3 to 65.3] | 39.3 [27.8 to 50.8]
Statistical Analysis 1: Comparison: Pemetrexed + Cisplatin; Hypothesis testing was done independently for each treatment arm (no direct treatment group comparison); Test type: Superiority or Other; 6-Month PFS Rate = 52.8, 95% CI 2-sided [40.3 to 65.3]
Statistical Analysis 2: Comparison: Pemetrexed + Carboplatin; Hypothesis testing was done independently for each treatment arm (no direct treatment group comparison); Test type: Superiority or Other; 6-Month PFS Rate = 39.3, 95% CI 2-sided [27.8 to 50.8]

2. Secondary Outcome: Overall Survival
Description: Defined as the time from randomization to the date of death from any cause.
Time Frame: Randomization to date of death from any cause (up to 1 year)
Population: Full Analysis Set: All patients randomized who received at least one dose of study drug
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Cisplatin | Pemetrexed + Carboplatin
Number analyzed (Participants) | 65 | 65
months | 11.7 [9.2 to 14.9] | 8.9 [6.0 to 12.2]

3. Secondary Outcome: Number of Participants With Tumor Response (as Basis for Response Rate)
Description: Best overall response was evaluated using RECIST Criteria which define when cancer patients improve ("respond"), stay the same ("stabilize"), or worsen ("progression") during treatment. CR: complete response, disappearance of all target lesions; PR: partial response, 30% decrease in sum of the longest diameter of target lesions; PD: progressive disease, 20% increase in sum of the longest diameter of target lesions; SD: stable disease, small changes not meeting above criteria. Response Rate: number of participants with response(CR+PR)per total population, multiplied by 100 to give a percentage.
Time Frame: Every 6 weeks for 6 months during the treatment period, and every 3 months during the follow-up period, until disease progression
Population: Full Analysis Set: All patients randomized who received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | Pemetrexed + Cisplatin | Pemetrexed + Carboplatin
Number analyzed (Participants) | 65 | 65
participants
  Partial Response | 21 | 13
  Stable Disease | 31 | 32
  Disease Progression | 7 | 15
  Unknown/Not Done | 6 | 5
Statistical Analysis 1: Comparison: Pemetrexed + Cisplatin; Response rates were evaluated separately for each treatment arm; Test type: Superiority or Other; Best Overall Response Rate (%) = 32.3, 95% CI [21.2 to 45.1]
Statistical Analysis 2: Comparison: Pemetrexed + Carboplatin; Response rates were evaluated separately for each treatment arm; Test type: Superiority or Other; Best Overall Response Rate (%) = 20.0, 95% CI [11.1 to 31.8]

4. Secondary Outcome: Time to Treatment Failure (TTF)
Description: Defined as time from randomization to the first date of disease progression, death due to any cause, or early discontinuation of treatment (any reason), whichever occurred first
Time Frame: Randomization to stopping of treatment, progression, death or initiation of further chemotherapy, whichever occurs first (up to 1 year)
Population: Full Analysis Set: All patients randomized who received at least one dose of study drug
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Cisplatin | Pemetrexed + Carboplatin
Number analyzed (Participants) | 65 | 65
months | 3.0 [2.3 to 4.6] | 3.4 [2.3 to 4.8]

5. Secondary Outcome: Pharmacology Toxicities
Description: Number of patients experiencing Grade 3 or 4 hematologic and non-hematologic adverse events (AEs) possibly related to study drug or protocol procedures in this study (a subset of those listed in the AE Module). AEs were graded using the Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0) for defining and grading specific adverse events. A grading (severity) scale is provided for each adverse event term. Grades range from 0 (none) to 5 (death). Grade 3 AEs are severe and undesirable; Grade 4 AEs are life-threatening or disabling.
Time Frame: Every 21-day cycle for up to 6 cycles
Population: Full Analysis Set: All patients randomized who received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | Pemetrexed + Cisplatin | Pemetrexed + Carboplatin
Number analyzed (Participants) | 65 | 65
participants
  Any Grade 3/4 Toxicity | 29 | 36
  Grade 3/4 Leucopenia | 8 | 12
  Grade 3/4 Neutropenia | 11 | 17
  Grade 3/4 Anemia | 5 | 7
  Grade 3/4 Thrombocytopenia | 2 | 11
  Grade 3/4 Nausea | 3 | 5
  Grade 3/4 Vomiting | 2 | 1
  Grade 3/4 Fatigue | 2 | 2
  Grade 3/4 Anorexia | 1 | 2
  Grade 3/4 Urinary Tract Infection | 0 | 2

ADVERSE EVENTS:
Arm/Group | Pemetrexed + Cisplatin | Pemetrexed + Carboplatin
Serious Adverse Events (participants affected / at risk) | 22/65 | 28/65
Other Adverse Events (participants affected / at risk) | 61/65 | 59/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Cisplatin (N=65) | Pemetrexed + Carboplatin (N=65)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 2 (2)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Chest pain (General disorders) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Performance status decreased (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Aspergillosis (Infections and infestations) | 0 (0) | 1 (1)
Cerebral fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 2 (3)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Mental disorder due to a general medical condition (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Cisplatin (N=65) | Pemetrexed + Carboplatin (N=65)
Anaemia (Blood and lymphatic system disorders) | 12 (13) | 19 (27)
Haemoglobinaemia (Blood and lymphatic system disorders) | 4 (4) | 12 (13)
Leukopenia (Blood and lymphatic system disorders) | 17 (27) | 24 (41)
Neutropenia (Blood and lymphatic system disorders) | 18 (27) | 25 (62)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (12) | 18 (39)
Conjunctivitis (Eye disorders) | 5 (5) | 2 (2)
Lacrimation increased (Eye disorders) | 6 (6) | 2 (2)
Constipation (Gastrointestinal disorders) | 17 (18) | 11 (13)
Diarrhoea (Gastrointestinal disorders) | 10 (12) | 10 (13)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 5 (5)
Nausea (Gastrointestinal disorders) | 42 (77) | 27 (46)
Stomatitis (Gastrointestinal disorders) | 5 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 24 (31) | 8 (10)
Fatigue (General disorders) | 25 (30) | 24 (31)
Mucosal inflammation (General disorders) | 5 (5) | 5 (9)
Oedema peripheral (General disorders) | 6 (6) | 3 (3)
Infection (Infections and infestations) | 6 (7) | 4 (5)
Rhinitis (Infections and infestations) | 2 (2) | 7 (7)
Alanine aminotransferase increased (Investigations) | 0 (0) | 4 (4)
Blood creatinine increased (Investigations) | 5 (5) | 2 (3)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 5 (5)
Weight decreased (Investigations) | 3 (3) | 8 (9)
Anorexia (Metabolism and nutrition disorders) | 16 (21) | 10 (12)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (5) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 4 (6)
Dizziness (Nervous system disorders) | 7 (9) | 3 (6)
Headache (Nervous system disorders) | 7 (9) | 5 (7)
Insomnia (Psychiatric disorders) | 5 (5) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 10 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6) | 6 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (6)
Rash (Skin and subcutaneous tissue disorders) | 3 (4) | 4 (7)
Hypertension (Vascular disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days